CLINICAL TRIAL: NCT04972968
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled, Dose-Ranging Study to Evaluate the Safety and Efficacy of ABBV-154 in Subjects With Polymyalgia Rheumatica (PMR) Dependent on Glucocorticoid Treatment
Brief Title: A Study to Evaluate the Change in Disease State and Adverse Events in Adult Participants With Polymyalgia Rheumatica (PMR) Dependent on Glucocorticoid Treatment, Receiving Subcutaneous Injections of ABBV-154
Acronym: AIM-PMR
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Strategic considerations
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: M20-370; 2021-000648-23 (EudraCT Number)
Record Dates: First submitted 2021-07-13; First posted 2021-07-22 (Actual); Results first posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Polymyalgia Rheumatica
Keywords: Polymyalgia Rheumatica; PMR; ABBV-154; Glucocorticoid
MeSH Terms: conditions — Polymyalgia Rheumatica | interventions — Glucocorticoids

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- ABBV-154 Dose A (Experimental): Participants in this group will receive dose A of ABBV-154 subcutaneously (SC) every other week (eow) for 52 weeks. In addition, participants will receive a glucocorticoid oral tablet taper.
  Interventions: Drug: ABBV-154; Drug: Glucocorticoid
- ABBV-154 Dose B (Experimental): Participants in this group will receive dose B of ABBV-154 SC eow for 52 weeks. In addition, participants will receive a glucocorticoid oral tablet taper.
  Interventions: Drug: ABBV-154; Drug: Glucocorticoid
- ABBV-154 Dose C (Experimental): Participants in this group will receive dose C of ABBV-154 SC eow for 52 weeks. In addition, participants will receive a glucocorticoid oral tablet taper.
  Interventions: Drug: ABBV-154; Drug: Glucocorticoid
- Placebo (Placebo Comparator): Participants will receive placebo SC eow for 52 weeks. In addition, participants will receive a glucocorticoid oral tablet taper.
  Interventions: Drug: Placebo; Drug: Glucocorticoid

INTERVENTIONS:
Drug: ABBV-154 — Subcutaneous Injection
  Arms: ABBV-154 Dose A; ABBV-154 Dose B; ABBV-154 Dose C
Drug: Placebo — Subcutaneous Injection
  Arms: Placebo
Drug: Glucocorticoid — Oral Tablet

SUMMARY:
Polymyalgia rheumatica (PMR) is an inflammatory disease causing shoulder, hip, and neck pain and stiffness, in adults aged 50 years or older. This study evaluates how safe and effective ABBV-154 is in participants with glucocorticoid-dependent PMR. Adverse events and change in disease activity will be assessed.

ABBV-154 is an investigational drug being evaluated for the treatment of PMR. Participants will be randomized into 1 of 4 treatment groups or arms, each arm receiving a different treatment. There is a 1 in 4 chance that a participant will be assigned to placebo. Around 160 participants, of at least 50 years of age, with PMR will be enrolled in the study at approximately 95 sites worldwide.

The study is compromised of a 52 week double-blind, placebo-controlled period and a follow-up visit 70 days after the last dose of the study drug. All participants will receive a glucocorticoid taper along with the assigned dose of ABBV-154 or placebo, subcutaneously (SC) every other week (eow).

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the study at a hospital or clinic. The effect of the treatment will be checked by medical assessments, blood tests, checking for side effects and completing questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Polymyalgia Rheumatica (PMR) and fulfillment of the 2012 European League Against Rheumatism/American College of Rheumatology (EULAR/ACR) provisional classification criteria for PMR.
* Must have had at least 2 episodes of unequivocal PMR flare.
* Must be on a stable dose of prednisone.
* Must be willing to follow the protocol-defined glucocorticoid tapering regimen.

Exclusion Criteria:

* Have been treated with a prior TNF antagonist.
* Current use of immunomodulators other than prednisone and hydroxychloroquine.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 181 (Actual)
Dates: Start 2021-09-09 (Actual); Primary Completion 2023-07-24 (Actual); Study Completion 2023-07-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (117):
- United States (31):
  - Arthritis and Rheumatism Associates /ID# 232089, Jonesboro, Arkansas
  - Providence Medical Foundation /ID# 228681, Fullerton, California
  - Care Access Research, Huntington Beach /ID# 228677, Huntington Beach, California
  - Purushotham & Akther Kotha MD, Inc /ID# 245391, La Mesa, California
  - Arthritis & Osteo Medical Ctr /ID# 228680, La Palma, California
  - Hans Richard Barthel, M.D., Inc /ID# 231902, Santa Barbara, California
  - Medvin Clinical Research /ID# 228675, Tujunga, California
  - Inland Rheum & Osteo Med Grp /ID# 228679, Upland, California
  - Denver Arthritis Clinic /ID# 245736, Denver, Colorado
  - Delaware Arthritis /ID# 230110, Lewes, Delaware
  - Arthritis & Rheumatic Disease Specialties /ID# 245448, Aventura, Florida
  - Rheumatology Associates of South Florida (RASF) - Clinical Research /ID# 232238, Boca Raton, Florida
  - International Medical Research /ID# 228765, Daytona Beach, Florida
  - Omega Research Debary, LLC /ID# 245450, DeBary, Florida
  - Lakes Research, LLC /ID# 228757, Miami, Florida
  - HMD Research LLC /ID# 228767, Orlando, Florida
  - Springfield Clinic /ID# 228840, Springfield, Illinois
  - Four Rivers Clinical Research /ID# 228858, Paducah, Kentucky
  - Rheumatology Consultants - Clinical Research /ID# 232137, Tupelo, Mississippi
  - Dartmouth-Hitchcock Medical Center /ID# 229557, Lebanon, New Hampshire
  - Ocean Rheumatology, PA /ID# 232539, Toms River, New Jersey
  - Hospital for Special Surgery /ID# 228577, New York, New York
  - St. Lawrence Health System /ID# 229702, Potsdam, New York
  - University of Rochester Medical Center /ID# 232554, Rochester, New York
  - Paramount Medical Research Con /ID# 228839, Middleburg Heights, Ohio
  - Clinical Research Source, Inc. /ID# 231903, Perrysburg, Ohio
  - Altoona Ctr Clinical Res /ID# 232493, Duncansville, Pennsylvania
  - Articularis Healthcare Group, Inc d/b/a Low Country Rheumatology /ID# 228860, Summerville, South Carolina
  - West Tennessee Research Institute /ID# 228854, Jackson, Tennessee
  - Rheumatology Care Center PLLC /ID# 232306, Bellaire, Texas
  - DM Clinical Research - Tomball /ID# 245512, Tomball, Texas
- Australia (8):
  - Emeritus Research Sydney /ID# 229166, Botany, New South Wales
  - Royal Prince Alfred Hospital /ID# 244888, Camperdown, New South Wales
  - BJC Health /ID# 244839, Paramatta, New South Wales
  - Tasman Health Care /ID# 230829, Southport, Queensland
  - The Queen Elizabeth Hospital /ID# 229049, Woodville South, South Australia
  - Emeritus Research /ID# 229270, Camberwell, Victoria
  - Austin Health /ID# 229164, Heidelberg, Victoria
  - Fiona Stanley Hospital /ID# 229050, Murdoch, Western Australia
- Rheuma-Zentrum Wien-Oberlaa GmbH /ID# 229436, Vienna, Vienna, Austria
- Canada (4):
  - Rheumatology Research Associates /ID# 230363, Edmonton, Alberta
  - The Waterside Clinic /ID# 230364, Barrie, Ontario
  - CISSSBSL -Hopital regional de Rimouski /ID# 228394, Rimouski, Quebec
  - Centre de Recherche Musculo-Squelettique /ID# 228392, Trois-Rivières, Quebec
- France (6):
  - CHU de Besancon - Jean Minjoz /ID# 244897, Besançon, Doubs
  - Hopital de la Cavale Blanche /ID# 228348, Brest, Finistere
  - CHU Montpellier - Hôpital Lapeyronie /ID# 228347, Montpellier, Herault
  - Centre Hospitalier du Mans /ID# 229044, Le Mans, Sarthe
  - CHRU Tours - Hopital Trousseau /ID# 228349, Chambray-lès-Tours
  - AP-HP - Hopital Cochin /ID# 231800, Paris
- Germany (5):
  - Medius Klinik Kirchheim /ID# 228660, Kirchheim unter Teck, Baden-Wurttemberg
  - Charite Universitaetsmedizin Berlin - Campus Mitte /ID# 228661, Berlin
  - Immanuel Krankenhaus Berlin /ID# 228659, Buch
  - MVZ Rheumatologie und Autoimmunmedizin Hamburg GmbH /ID# 228658, Hamburg
  - Rheumazentrum Ratingen /ID# 245183, Ratingen
- Hungary (9):
  - Debreceni Egyetem Klinikai Kozpont /ID# 241674, Debrecen, Hajdú-Bihar
  - Obudai Egeszsegugyi Centrum Kft. Zalaegerszeg /ID# 229759, Zalaegerszeg, Zala County
  - Clinexpert Kft /ID# 229677, Budapest
  - Obudai Egeszsegugyi Centrum Kft. /ID# 231121, Budapest
  - Bekes Megyei Kozponti Korhaz Pandy Kalman Tagkorhaz /ID# 229758, Gyula
  - Kistarcsai Flor Ferenc Korhaz /ID# 229676, Kistarcsa
  - Csongrad-Csanad Megyei Dr. Bugyi Istvan Korhaz /ID# 229793, Szentes
  - CMED Rehabilitacios es Diagnosztikai Kozpont /ID# 230065, Székesfehérvár
  - Vital Medical Center Orvosi es Fogaszati Kozpont (Vital Medicina Kft.) /ID# 229674, Veszprém
- Italy (6):
  - ASL 3 Genovese - Ospedale la Colletta /ID# 229282, Arenzano, Genova
  - A.O.U. Citta della Salute e della Scienza di Torino /ID# 229080, Turin, Torino
  - Azienda Ospedaliero-Universitaria di Modena /ID# 228825, Modena
  - Fondazione IRCCS Policlinico /ID# 245274, Pavia
  - Azienda Ospedaliero-Universitaria Senese-Ospedale Santa Maria delle Scotte /ID# 245273, Siena
  - Azienda Ospedaliera Universitaria Friuli Centrale/Presidio Ospedaliero Universit /ID# 228815, Udine
- Japan (12):
  - Daido Clinic /ID# 230204, Nagoya, Aichi-ken
  - NHO Nagoya Medical Center /ID# 232420, Nagoya, Aichi-ken
  - National Hospital Organization Shimoshizu National Hospital /ID# 230500, Yotsukaido-shi, Chiba
  - Matsuyama Red Cross Hospital /ID# 230458, Matsuyama, Ehime
  - Sanuki Municipal Hospital /ID# 230202, Sanuki-shi, Kagawa-ken
  - Kuwana city medical center /ID# 231936, Kuwana-shi, Mie-ken
  - Kyushu University Beppu Hospital /ID# 232250, Beppu-shi, Oita Prefecture
  - Japanese Red Cross Okayama Hospital /ID# 230857, Okayama, Okayama-ken
  - Rinku Hashimoto Rheumatology Orthopaedics /ID# 246532, Izumisano, Osaka
  - Osaka Medical and Pharmaceutical University Hospital /ID# 246530, Takatsuki-shi, Osaka
  - Tokyo Medical And Dental University Hospital /ID# 232206, Bunkyo-ku, Tokyo
  - Toyama Prefectural Central Hospital /ID# 230616, Toyama, Toyama
- Netherlands (5):
  - ZiekenhuisGroep Twente /ID# 229071, Almelo
  - Universitair Medisch Centrum Groningen /ID# 227727, Groningen
  - Medisch Centrum Leeuwarden /ID# 245442, Leeuwarden
  - Maastricht Universitair Medisch Centrum /ID# 227779, Maastricht
  - Maasstad Ziekenhuis /ID# 228064, Rotterdam
- New Zealand (6):
  - Optimal Clinical Trials Ltd /ID# 229048, Grafotn, Auckland
  - Aotearoa Clinical Trials /ID# 229099, Papatoetoe, Auckland
  - Timaru Medical Specialists Ltd /ID# 229098, Timaru, Canterbury
  - Waikato Hospital /ID# 229047, Hamilton, Waikato Region
  - Wellington Regional Hospital /ID# 229490, Newtown, Wellington Region
  - CGM Research Trust /ID# 244893, Christchurch Central
- Poland (6):
  - AI Centrum Medyczne Sp. z o.o. sp.k. /ID# 228951, Poznan, Greater Poland Voivodeship
  - Ortopedyczno-Rehabilitacyjny Szpital Kliniczny im. Wiktora Degi /ID# 228314, Poznan, Greater Poland Voivodeship
  - Szpital Uniwersytecki nr 2 im. dr. Jana Biziela /ID# 228353, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Niepubliczny Zaklad Opieki Zdrowotnej Biogenes Sp. z o.o /ID# 228357, Wroclaw, Lower Silesian Voivodeship
  - Centrum Medyczne Reuma Park /ID# 244813, Warsaw, Masovian Voivodeship
  - Nova Reuma Domyslawska I Rusilowicz - Spolka Partnerska Lekarza Reumatologa I Fi /Id# 228466, Bialystok, Podlaskie Voivodeship
- South Korea (2):
  - Hanyang University Seoul Hospital /ID# 228719, Seoul, Seoul Teugbyeolsi
  - Kyungpook National University Hospital /ID# 228716, Daegu
- Spain (7):
  - Hospital Clínico Universitario de Santiago-CHUS /ID# 244868, Santiago de Compostela, A Coruna
  - Consorci Corporacio Sanitaria Parc Tauli Sabadell /ID# 244866, Sabadell, Barcelona
  - Hospital Universitario Marques de Valdecilla /ID# 229297, Santander, Cantabria
  - Hospital Universitario Canarias /ID# 229451, San Cristóbal de La Laguna, Santa Cruz De Tenerife
  - Hospital Clinic de Barcelona /ID# 229295, Barcelona
  - Hospital General Universitario Gregorio Maranon /ID# 229302, Madrid
  - Hospital Clinico Universitario San Carlos /ID# 229296, Madrid
- United Kingdom (9):
  - North West Anglia NHS Foundation Trust /ID# 230866, Bretton, Cambridgeshire
  - Leicester Royal Infirmary /ID# 231967, Leicester, England
  - The Royal Free London NHS Foundation Trust /ID# 231707, London, London, City of
  - Norfolk and Norwich University Hospitals NHS Foundation Trust /ID# 231966, Norwich, Norfolk
  - Cardiff & Vale University Health Board /ID# 245297, Cardiff, Wales
  - UH Coventry & Warwickshire /ID# 228588, Coventry
  - NHS Lothian /ID# 245293, Edinburgh
  - Liverpool University Hospitals NHS Foundation Trust /ID# 245296, Liverpool
  - Portsmouth Hospitals University NHS Trust /ID# 245291, Portsmouth

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols, analyses plans, clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous independent scientific research, and will be provided following review and approval of a research proposal and statistical analysis plan and execution of a data sharing statement. Data requests can be submitted at any time after approval in the US and/or EU and a primary manuscript is accepted for publication. For more information on the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: In this Double-Blind study, 181 glucocorticoid dependent PMR subjects were randomized into 4 groups and dosed for 52 weeks. Subjects were dosed SC: Placebo, ABBV-154 (40mg,150mg, or 340mg) with a glucocorticoid taper EOW. Beginning at Week 3, subjects were to taper prednisone/prednisolone per the protocol-defined glucocorticoid taper schedule to 0mg prednisone equivalent by Week 24.
Groups:
- ABBV-154, 40mg SC: Participants in this group received 40mg dose of ABBV-154 SC eow for 52 weeks. In addition, participants received a glucocorticoid oral tablet taper.
  ABBV-154: 40mg SC
  Glucocorticoid: Oral Tablet
- ABBV-154, 150mg SC: Participants in this group received 150mg dose of ABBV-154 SC eow for 52 weeks. In addition, participants received a glucocorticoid oral tablet taper.
  ABBV-154: 150mg SC
  Glucocorticoid: Oral Tablet
- ABBV-154, 340mg SC: Participants in this group received 340mg dose of ABBV-154 SC eow for 52 weeks. In addition, participants received a glucocorticoid oral tablet taper.
  ABBV-154: 340mg SC
  Glucocorticoid: Oral Tablet
Period: Overall Study
Arm/Group | Placebo | ABBV-154, 40mg SC | ABBV-154, 150mg SC | ABBV-154, 340mg SC
Started | 50 | 42 | 45 | 44
Completed | 12 | 8 | 8 | 7
Not Completed | 38 | 34 | 37 | 37
Not completed — Adverse Event | 3 | 1 | 1 | 7
Not completed — Lack of Efficacy | 2 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 7 | 4 | 3 | 2
Not completed — Study Terminated by Sponsor | 25 | 28 | 32 | 27
Not completed — Other | 1 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Participants received placebo subcutaneously (SC) every other week (eow) for 52 weeks. In addition, participants received a glucocorticoid oral tablet taper.
  Placebo: Subcutaneous Injection Glucocorticoid: Oral Tablet
- ABBV-154 40mg SC: Participants in this group received 40mg dose of ABBV-154 SC eow for 52 weeks. In addition, participants received a glucocorticoid oral tablet taper.
  ABBV-154: Subcutaneous Injection Glucocorticoid: Oral Tablet
- ABBV-154 150mg SC: Participants in this group received 150mg dose of ABBV-154 SC eow for 52 weeks. In addition, participants received a glucocorticoid oral tablet taper.
  ABBV-154: Subcutaneous Injection Glucocorticoid: Oral Tablet
- ABBV-154 340mg SC: Participants in this group received 340mg dose of ABBV-154 SC eow for 52 weeks. In addition, participants received a glucocorticoid oral tablet taper.
  ABBV-154: Subcutaneous Injection Glucocorticoid: Oral Tablet
- Total: Total of all reporting groups
Arm/Group | Placebo | ABBV-154 40mg SC | ABBV-154 150mg SC | ABBV-154 340mg SC | Total
Number analyzed (Participants) | 50 | 42 | 45 | 44 | 181
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.0 (7.15) | 67.5 (7.98) | 69.8 (8.34) | 69.1 (6.23) | 69.4 (7.50)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 30 | 25 | 29 | 117
  Male | 17 | 12 | 20 | 15 | 64
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 2 | 2 | 5
  Not Hispanic or Latino | 49 | 42 | 43 | 42 | 176
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Baseline Glucocorticoid Dose (mg/day) [Least Squares Mean (Standard Deviation); unit: mg/day] | 9.21 (3.801) | 9.45 (3.378) | 9.10 (3.519) | 9.52 (3.317) | 9.31 (3.495)

OUTCOME MEASURES:

1. Primary Outcome: Time to Flare
Description: Flare is defined as, presence of clinical signs and symptoms of PMR and requirement to increase the glucocorticoid dose per investigator.
Time Frame: From first dose of study drug to Week 52
Population: ITT Population
Measure: Median (95% Confidence Interval); unit: days
Groups:
- Placebo: Participants will receive placebo SC EOW for 24 weeks. In addition, participants will receive a glucocorticoid oral tablet taper.
  Placebo: Subcutaneous Injection
  Glucocorticoid: Oral Tablet
- ABBV-154, 40mg SC: Participants in this group received 40mg dose of ABBV-154 SC EOW for 24 weeks. In addition, participants received a glucocorticoid oral tablet taper.
  ABBV-154: 40mg SC
  Glucocorticoid: Oral Tablet
- ABBV-154, 150mg SC: Participants in this group received 150mg dose of ABBV-154 SC EOW for 24 weeks. In addition, participants received a glucocorticoid oral tablet taper.
  ABBV-154: 150mg SC
  Glucocorticoid: Oral Tablet
- ABBV-154, 340mg SC: Participants in this group received 340mg dose of ABBV-154 SC EOW for 24 weeks. In addition, participants received a glucocorticoid oral tablet taper.
  ABBV-154: 340mg SC
  Glucocorticoid: Oral Tablet
Arm/Group | Placebo | ABBV-154, 40mg SC | ABBV-154, 150mg SC | ABBV-154, 340mg SC
Number analyzed (Participants) | 50 | 42 | 45 | 44
days | 113 [84 to 141] | 225 [140 to NA] — Not calculable/estimable due to low number of participants with flares | NA [141 to NA] — Not calculable/estimable due to low number of participants with flares | NA [NA to NA] — Not calculable/estimable due to low number of participants with flares
Statistical Analysis 1: Comparison: Placebo vs ABBV-154, 40mg SC; Test type: Superiority; p = 0.012, Log Rank — P-value <= 0.05; Stratified by baseline randomization stratification factors [Glucocorticoid use at Baseline (>= 10 mg/day; < 10 mg/day prednisone equivalent)]; Cox Proportional Hazard = 0.490, 95% CI 2-sided [0.273 to 0.878]
Statistical Analysis 2: Comparison: Placebo vs ABBV-154, 150mg SC; Test type: Superiority; p = 0.004, Log Rank — P-value <= 0.01; [statistical method as in outcome 1, analysis 1]; Cox Proportional Hazard = 0.443, 95% CI 2-sided [0.248 to 0.794]
Statistical Analysis 3: Comparison: Placebo vs ABBV-154, 340mg SC; Test type: Superiority; p < 0.001, Log Rank — P-value <= 0.001; [statistical method as in outcome 1, analysis 1]; Cox Proportional Hazard = 0.198, 95% CI 2-sided [0.094 to 0.419]

2. Secondary Outcome: Percentage of Participants Achieving Flare-Free State
Description: Percentage of participants achieving flare-free state.
Time Frame: Up to Week 24
Population: ITT Population with data available for analysis
Measure: Number; unit: percentage of participants
Groups:
- Placebo: Participants received placebo subcutaneously (SC) every other week (eow) for 52 weeks. In addition, participants received a glucocorticoid oral tablet taper.
- ABBV-154 40mg SC: Participants in this group received 40mg dose of ABBV-154 SC eow for 52 weeks. In addition, participants received a glucocorticoid oral tablet taper.
- ABBV-154 150mg SC: Participants in this group received 150mg dose of ABBV-154 SC eow for 52 weeks. In addition, participants received a glucocorticoid oral tablet taper.
- ABBV-154 340mg SC: Participants in this group received 340mg dose of ABBV-154 SC eow for 52 weeks. In addition, participants received a glucocorticoid oral tablet taper.
Arm/Group | Placebo | ABBV-154 40mg SC | ABBV-154 150mg SC | ABBV-154 340mg SC
Number analyzed (Participants) | 39 | 28 | 32 | 34
percentage of participants | 11 | 13 | 15 | 24
Statistical Analysis 1: Comparison: Placebo vs ABBV-154 40mg SC; Test type: Superiority; p = 0.107, Cochran-Mantel-Haenszel; Mean Difference (Net) = 18.7, 95% CI 2-sided [-4.0 to 41.4] — From Cochran-Mantel-Haenszel test adjusting for baseline randomization stratification factors [Glucocorticoid (GC) use at baseline (≥ 10 mg/day; < 10 mg/day prednisone equivalent); Length of prior GC treatment for PMR (≤ 1 year; > 1 year)]
Statistical Analysis 2: Comparison: Placebo vs ABBV-154 150mg SC; Test type: Superiority; p = 0.092, Cochran-Mantel-Haenszel — P-value ≤ 0.1; Mean Difference (Net) = 18.9, 95% CI 2-sided [-3.1 to 41.0] — Cochran-Mantel-Haenszel test adjusting for baseline randomization stratification factors [Glucocorticoid use at baseline (≥ 10 mg/day; < 10 mg/day prednisone equivalent); Length of prior GC treatment for PMR (≤ 1 year; > 1 year)]
Statistical Analysis 3: Comparison: Placebo vs ABBV-154 340mg SC; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — P-value ≤ 0.001; Mean Difference (Net) = 41.9, 95% CI 2-sided [21.4 to 62.3] — [estimate comment as in outcome 2, analysis 2]

3. Secondary Outcome: Cumulative Glucocorticoid Dose
Description: Cumulative glucocorticoid dose.
Time Frame: Week 24
Population: ITT Population with data available for analysis
Measure: Mean (Standard Deviation); unit: Glucocorticoid dose (mg)
Arm/Group | Placebo | ABBV-154 40mg SC | ABBV-154 150mg SC | ABBV-154 340mg SC
Number analyzed (Participants) | 36 | 28 | 29 | 30
Glucocorticoid dose (mg) | 984.576 (524.6579) | 823.411 (397.9403) | 734.310 (332.3137) | 759.450 (381.1683)
Statistical Analysis 1: Comparison: Placebo vs ABBV-154 40mg SC; Test type: Superiority; p = 0.144, ANCOVA; P-value based on an Analysis of covariance (ANCOVA) model adjusting for baseline randomization stratification factors; Mean Difference (Net) = -88.67, 95% CI 2-sided [-208.04 to 30.71] — 95% CI based on an Analysis of covariance (ANCOVA) model adjusting for baseline randomization stratification factors [GC use at baseline (≥ 10 mg/day; < 10 mg/day prednisone equivalent);
Statistical Analysis 2: Comparison: Placebo vs ABBV-154 150mg SC; Test type: Superiority; p = 0.007, ANCOVA — P-value ≤ 0.01; Mean Difference (Net) = -164.76, 95% CI 2-sided [-283.62 to -45.89] — P-value and 95% CI are based on an Analysis of covariance (ANCOVA) model adjusting for baseline randomization stratification factors [Glucocorticoid use at baseline (≥ 10 mg/day; < 10 mg/day prednisone] equivalent);
Statistical Analysis 3: Comparison: Placebo vs ABBV-154 340mg SC; Test type: Superiority; p = 0.003, ANCOVA — P-value ≤ 0.01; Mean Difference (Final Values) = -182.55, 95% CI 2-sided [-300.52 to -64.58] — P-value and 95% CI based on an Analysis of covariance (ANCOVA) model adjusting for baseline randomization stratification factors [Glucocorticoid use at baseline (≥ 10 mg/day; < 10 mg/day prednisone equivalent)

4. Secondary Outcome: Change From Baseline in Glucocorticoid Dose
Description: Change from Baseline in glucocorticoid dose.
Time Frame: Week 24
Population: ITT Population with data available for analysis
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Placebo | ABBV-154 40mg SC | ABBV-154 150mg SC | ABBV-154 340mg SC
Number analyzed (Participants) | 36 | 28 | 29 | 30
mg | -4.96 (3.943) | -6.29 (3.384) | -7.40 (3.554) | -7.88 (3.398)
Statistical Analysis 1: Comparison: Placebo vs ABBV-154 40mg SC; Test type: Superiority; p = 0.039, ANCOVA — P-value <= 0.05; P-value based on ANCOVA adjusting for baseline randomization stratification factors (GC use at baseline); Mean Difference (Net) = -1.58, 95% CI 2-sided [-3.08 to -0.08]
Statistical Analysis 2: Comparison: Placebo vs ABBV-154 150mg SC; Test type: Superiority; p < 0.001, ANCOVA — P-value <= 0.001; P-value based on an ANCOVA model adjusting for baseline randomization stratification factors (GC use at baseline); Mean Difference (Final Values) = -2.66, 95% CI 2-sided [-4.15 to -1.16] — 95% CI based on an ANCOVA model adjusting for baseline randomization stratification factors (GC use at baseline)
Statistical Analysis 3: Comparison: Placebo vs ABBV-154 340mg SC; Test type: Superiority; p < 0.001, ANCOVA — P-value <= 0.001; P-value based on an ANCOVA model adjusting for baseline randomization stratification factors (GC use at baseline); Mean Difference (Final Values) = -3.00, 95% CI 2-sided [-4.49 to -1.52] — 95% CI based on an ANCOVA model adjusting for baseline randomization stratification factors (GC use at baseline)

ADVERSE EVENTS:
Time Frame: All-cause mortality were reported from enrollment to the end of study, median time on follow up was 288.5, 292.0, 300.0, and 299.0 Days for Placebo and ABBV-154 (40mg/150mg/340mg), respectively. Treatment-emergent adverse events and serious adverse events were collected from first dose of study drug within 70 days after the last dose of study drug; mean duration on study drug was 235.2, 239.9, 234.6 and 230.3 days for Placebo and ABBV-154 (40mg/150mg/340mg), respectively.
Arm/Group | Placebo | ABBV-154 40mg SC | ABBV-154 150mg SC | ABBV-154 340mg SC
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/42 | 0/45 | 0/44
Serious Adverse Events (participants affected / at risk) | 8/50 | 5/42 | 8/45 | 9/44
Other Adverse Events (participants affected / at risk) | 27/50 | 25/42 | 30/45 | 37/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=50) | ABBV-154 40mg SC (N=42) | ABBV-154 150mg SC (N=45) | ABBV-154 340mg SC (N=44)
ATRIAL FIBRILLATION (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
CORONARY ARTERY DISEASE (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
LEFT VENTRICULAR FAILURE (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SUPRAVENTRICULAR TACHYCARDIA (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
VENTRICULAR EXTRASYSTOLES (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ATRIAL SEPTAL DEFECT (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
INGUINAL HERNIA (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PANCREATIC PSEUDOCYST (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PANCREATITIS (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CHOLANGITIS ACUTE (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
APPENDICITIS PERFORATED (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CELLULITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PERITONITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PNEUMONIA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
PNEUMONIA PNEUMOCOCCAL (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
SEPSIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
UROSEPSIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
DEHYDRATION (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
DIABETES MELLITUS (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
ACUTE MYELOID LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PROSTATE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
DIZZINESS (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SCIATICA (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
THALAMIC INFARCTION (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
FEMALE GENITAL TRACT FISTULA (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
DYSPNOEA AT REST (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=50) | ABBV-154 40mg SC (N=42) | ABBV-154 150mg SC (N=45) | ABBV-154 340mg SC (N=44)
NEUTROPENIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 3 (4) | 0 (0)
DIARRHOEA (Gastrointestinal disorders) | 4 (4) | 2 (3) | 2 (2) | 3 (4)
NAUSEA (Gastrointestinal disorders) | 2 (3) | 3 (3) | 2 (2) | 3 (4)
FATIGUE (General disorders) | 2 (2) | 3 (3) | 4 (5) | 2 (2)
INJECTION SITE ERYTHEMA (General disorders) | 0 (0) | 2 (3) | 3 (4) | 2 (5)
INJECTION SITE PAIN (General disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
INJECTION SITE RASH (General disorders) | 0 (0) | 1 (2) | 3 (7) | 1 (1)
OEDEMA PERIPHERAL (General disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
PYREXIA (General disorders) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 9 (9) | 9 (9) | 5 (5) | 7 (7)
NASOPHARYNGITIS (Infections and infestations) | 3 (4) | 4 (5) | 4 (5) | 7 (9)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 2 (2) | 2 (3) | 3 (3) | 2 (2)
URINARY TRACT INFECTION (Infections and infestations) | 5 (9) | 3 (3) | 2 (5) | 6 (9)
CONTUSION (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 2 (2) | 3 (7)
SKIN LACERATION (Injury, poisoning and procedural complications) | 0 (0) | 3 (5) | 1 (1) | 2 (2)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 3 (5) | 4 (4) | 6 (6) | 3 (5)
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 3 (3) | 0 (0)
ROTATOR CUFF SYNDROME (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2) | 3 (4) | 1 (1)
DIZZINESS (Nervous system disorders) | 3 (3) | 0 (0) | 1 (1) | 2 (2)
HEADACHE (Nervous system disorders) | 2 (2) | 3 (3) | 4 (4) | 5 (10)
COUGH (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 4 (4)
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (4) | 1 (1) | 0 (0)
RASH (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2) | 2 (2) | 3 (3)
HYPERTENSION (Vascular disorders) | 5 (5) | 1 (1) | 4 (4) | 3 (3)

LIMITATIONS AND CAVEATS:
AbbVie has decided to discontinue further subject enrollment in the M20-370 (ABBV-154) study. This decision is not based on a safety or an efficacy signal; rather this decision was made because of a change in AbbVie's development.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-02-21): https://cdn.clinicaltrials.gov/large-docs/68/NCT04972968/Prot_000.pdf
  • Statistical Analysis Plan (2022-08-03): https://cdn.clinicaltrials.gov/large-docs/68/NCT04972968/SAP_001.pdf